CLINICAL TRIAL: NCT06253819
Title: Investigation of Respiratory Functions, Exercise Endurance and Functional Capacity in Geriatric Individuals With Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Alper Kemal Gürbüz, Research Asistant at physiotherapy and rehabilitation department, Kırıkkale University
Other Study IDs: Gurbuz05
Record Dates: First submitted 2024-01-07; First posted 2024-02-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome; Respiratory Disease; Exercise Capacity; Respiratory Muscle
MeSH Terms: conditions — Metabolic Syndrome; Respiration Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- geriatrics individuals with metabolic syndrome
  Interventions: Other: survey and physical test
- geriatrics individuals without metabolic syndrome
  Interventions: Other: survey and physical test

INTERVENTIONS:
Other: survey and physical test — 6 min. walking test respiratory function test 30 second sit-stand test respiratory muscle test tıme up and go corbin posture analysis Waist/Hip Circumference Ratio Glucose and Cholesterol values Lanss Neuropathic Pain Scale

SUMMARY:
Metabolic syndrome (MetS) or syndrome X, which is increasingly prevalent in the world and in our country, is a disease that includes abdominal obesity, dyslipidaemia, impaired glycaemic control and hypertension components. It causes cardiovascular events such as myocardial hypertrophy, left ventricular diastolic dysfunction, atrial dilatation and atrial fibrillation. Low physical activity level may be caused by various factors such as environmental and genetic factors, age, race, sarcopenia, poor eating habits, postmenopausal period and smoking history. It has been reported that factors such as genetic differences, diet, physical activity, age, gender and eating habits affect the prevalence of (MetS) and its components. Metabolic syndrome is a fatal endocrinopathy that starts with insulin resistance and is accompanied by systemic disorders such as abdominal obesity, glucose intolerance or diabetes mellitus, dyslipidaemia, hypertension and coronary artery disease (CAD). Although the prevalence of metabolic syndrome, which is accepted as an important public health problem in both developed and developing countries, varies according to different geographical and ethnic characteristics, definitions used, age and gender characteristics of populations, it shows a global increase and is considered as a pandemic affecting 20% to 30% of the adult population in many countries. The likelihood of metabolic syndrome increases in geriatric individuals due to some changes caused by aging. In a study conducted in geriatric individuals in our country, the incidence of metabolic syndrome was reported as 36.0%.

As a result of ageing, degenerative changes in the central and peripheral vestibular system have been found. With age, the ability to regulate movement is impaired as a result of insufficient information in any of the sensory receptors or any disorder affecting the processing of these messages. This directly affects functional capacity. In elderly individuals, tolerance to physical effort decreases due to a decrease in maximal oxygen consumption and maximal heart rate. Systolic and diastolic blood pressure increases. The number of respirations per minute increases in the elderly due to the difficulty in chest cage adaptation.Aging causes a decrease in the elasticity of the lung. The respiratory surface area, which is up to 75 square metres (m²) in young adults (due to damage to the inter-alveolar septum during aging), decreases by approximately 3 m² per decade. Systematic changes seen with aging also have negative effects on functional status and exercise endurance.

In sarcopenia, which is defined as a decrease in muscle mass and strength with advancing age, there is an irreversible decrease in the number of muscle fibres and myofibrils contained in each muscle fibre. From the age of 20 years to 70 years, approximately 40% loss in muscle mass and 30-50% decrease in muscle strength occur. It is stated that this loss starts at the age of 25, but muscle mass and muscle strength are lost at a rate of 1% per year from the age of 50.

In geriatric rehabilitation, patients' functionality, balance and fall problems have an important place. On the other hand, cardiac risk is increased in geriatric individuals and respiratory assessments have an important place. Metabolic syndrome is 7 times more common in individuals with maximal oxygen consumption (VO2 max) below 29 mL-kg-1 -min-1 than in those with VO2 max above 35.5 mL-kg-1 -min-1. Metabolic syndrome directly affects the pulmonary system.

In the light of the results obtained from the studies in the literature, degenerative changes are observed in many systems in geriatric individuals and while the incidence of metabolic syndrome in these individuals is high, the number of studies evaluating their effects is not sufficient. Based on these deficiencies, it is aimed to reveal the effects of respiratory muscle strength, pulmonary function, exercise endurance and functional level in geriatric individuals with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* To be able to communicate verbally
* Being able to walk independently
* To be able to read and write
* Volunteering to participate in the study

Exclusion Criteria:

* Mini Mental Status Scale less than 24
* Presence of orthopaedic condition preventing physical activity
* Having undergone cardiovascular surgery
* Having a pacemaker

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: In Kırıkkale Merkez Hürriyet Family Health Centre, all elderly individuals aged 65 years and over who meet the inclusion and exclusion criteria and who volunteered to participate in the study will be collected by face-to-face interview method using evaluation forms.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
functional status | 3 minute
  30 second sit-stand test: The patient is asked to sit up and down as quickly as possible in a chair with a seat height of 43.2 cm and a supported back. The patient sits on the chair. He crosses his hands on his chest. 2 attempts are made before the test. The duration of 30 seconds is kept with a stopwatch and the number of sit-ups is noted. Less than 10 sit-ups in 30 seconds indicates lower extremity muscle weakness.
balance and function | 2 minute
  Time up go, The individual is asked to get up from the chair without using his/her hands and walk 3 metres at a normal walking speed, then turn around and walk back to the chair and sit down.

SECONDARY OUTCOMES:
respiratory function | 5 minute
  Assessment of pulmonary function of individuals respiratory The function test is performed in a seated position with the shoulders relaxed in a chair without armrests, with back support, using the device. Lung volumes (FEV1/FVC) from the pulmonary function test are recorded.
respiratory muscle strenght | 2 minute
  Respiratory muscle strength will be measured non-invasively. A respiratory muscle strength measuring device (Power Breathe International Ltd, UK) will be used for the assessment. For the assessment, the athletes were placed in a seated position in a back-supported chair without armrests, with shoulders relaxed and using a nose clip. The athletes were asked to take a deep breath through the device placed in the mouth and the maximum inspiratory pressure (cmH2O) obtained was recorded. The assessment was repeated 3 times and mean values were recorded.
Quality of life, questionnaire questions on quality of life | 2 minute
  Barthel index,The Barthel Index is a detailed, unbiased, easily applicable, understandable scale that investigates the cause-effect relationship and evaluates all steps of activities of daily living. According to the Barthel Index, patients are evaluated as 0-20 points fully dependent, 21-61 points highly dependent, 62- 90 moderately dependent, 91-99 points mildly dependent and 100 points fully independent. In studies in which the Barthel Index was used, 60 points were taken as the limit and scores above 60 explain the ability to function independently.
pain level | 5 minute
  Lanss Neuropathic Pain Scale, The pain scale is a simple but useful bedside test for the differential diagnosis of neuropathic pain and nociceptive pain. The LANSS consists of two parts; the first part, which is completed by the patient and the second part, which includes a brief physical examination by the physician. Five self-answered questions (maximum score 16 points) describe experiences associated with neuropathic pain (such as pins and needles, paresthesia, skin discolouration due to autonomic changes, electrification and burning pain). In the physical examination part (maximum score), the presence of allodynia is tested by touching the painful and non-painful area with cotton wool. If the score is 12 and above, it is classified as neuropathic pain, and if the score is below 12, it is classified as nociceptive pain.
functional exercise capacity | 10 minute
  6 min walk test, The 6-minute walk test has good reproducibility and correlation with other functional capacity measurements. The walking distance of a normal person in 6 minutes is 400-700m. A 30 metre track is set up. The patient is brought to the starting line. The patient is informed that he/she should walk on the track at his/her own walking pace for 6 minutes, that he/she can stop the test at any time if he/she has a complaint, that he/she can stop and rest if he/she needs during the test and that he/she should continue the test until the command "test is over" is given. And the stopwatch is started and the test is started with the command "test started" and the test is terminated with the command "test over". During the test, if the patient stops and rests and takes a break from the test, the stopwatch is not stopped.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No